CLINICAL TRIAL: NCT02532959
Title: Pilot Study to Evaluate Diagnostic Breath Analysis for Early Detection of Systemic Inflammatory Response Syndrome (SIRS) and Sepsis
Brief Title: Diagnostic Breath Analysis Study to Detect Sepsis
Status: Completed | Type: Observational
Sponsor: Landon Pediatric Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Study:177
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Puerperal: [Major Infection] or [Sepsis]
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath saved for re-test in thirty days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic Breath Analysis: Patients at risk of SIRS
  Interventions: Device: Diagnostic Breath Analysis

INTERVENTIONS:
Device: Diagnostic Breath Analysis — Conduct exhaled breath samples

SUMMARY:
Analysis of exhaled breath samples using a high-speed gas chromatography medical device will identify Volatile Organic Compounds (VOC) that are specifically associated with SIRS and Sepsis.

Primary outcome measures will include the assessment of the zNose Diagnostic Breath Analysis System, which includes high-speed gas chromatography, in the early detection of SIRS and Sepsis as compared with current SIRS and Sepsis evaluation methods.

DETAILED DESCRIPTION:
Exhaled breath samples were collected in a Tedlar bag or with a proprietary collection tube. The collection devices are clean and intended for single-use. They are manufactured with approved medical grade materials. Patients were asked to breath into a single-use, medical grade mouthpiece which is connected to the collection bag or tube. The design of the collection devices does not allow the patient to rebreathe the exhaled gas sample. Patients enrolled in the clinical study were asked to breathe into the breath collection device for 2 to 4 breaths. Breath collection is completely non-invasive. Breath samples were held for 30 days and retested at the end of the 30 day period to determine if the VOC profile has changed over time.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Age 18 years of age or older
2. Able to give written and dated informed consent prior to any study specific procedures.
3. Able to follow instructions for specific breathing maneuvers.
4. Able to breath into a medical grade tube, vial or bag.
5. Initial assessment and screening indicates SIRS or Sepsis.

Exclusion Criteria:

Exclusion Criteria

1. Cognitively impaired and unable to complete informed consent documents.
2. Unable to follow instructions during testing.
3. Severe dyspnea.
4. Use of supplement oxygen which cannot be discontinued during testing.
5. Unable to perform breathing maneuvers required to provide multiple breath samples.
6. Swallowing disorders or chronic aspiration.
7. History of pneumothorax.
8. Patients requiring mechanical ventilation
9. Patients who are pregnant.
10. Patients who have smoked cigarettes or cigars within 30 days prior to trial admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients enter through Emergency Room, are identified at risk for SIRS
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic Breath Analysis | 6 months
  Diagnostic Breath Analysis to identify Volatile Organic Compounds (VOC) associated with Sepsis and SIRS

CONTACTS AND LOCATIONS:
Overall Officials: Crhis Landon, MD, Principal Investigator — Ventura County Medical Center
Locations (1):
- Ventura County Medical Center, Ventura, California, United States